CLINICAL TRIAL: NCT01182298
Title: Study to Evaluate the Genetic, Epigenetic, and Proteomic Expression in Latino Participants With and Without HIV Coinfection Receiving Treatment for Hepatitis C
Brief Title: Open Label Study to Evaluate Chronic Hepatitis C Treatment in Latino Subjects With and Without HIV Co-infection
Acronym: LATHCV
Status: Terminated | Type: Observational
Why Stopped: small number of patients enrolled
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: FDI Clinical Research (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100159; 10-I-0159 (Registry Identifier: CLINICAL TRIALS)
Record Dates: First submitted 2010-08-13; First posted 2010-08-16 (Estimated); Results first posted 2014-10-02 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2014-09

CONDITIONS: Hepatitis C; HIV
Keywords: Latino; HCV; pegIFN; Viral Kinetics; IL-28 Haplotype
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and serum storage.

GROUPS / COHORTS (1):
- Hepatitis C: latino participants with Hepatitis C

SUMMARY:
* Peginterferon alfa-2a has been approved by the U.S. Food and Drug Administration (FDA) to treat adults with chronic hepatitis C virus (HCV) infection with liver disease who have not been previously treated with interferon-alpha drugs (which improve immune system response to infection). Ribavirin has been approved by the FDA and is usually given in combination with interferon drugs such as peginterferon alfa-2a for treatment of chronic HCV.
* Recent research shows that Latino whites do not respond as well to treatment with peginterferon alfa-2a and ribavirin as non-Latino whites. Various factors such as excessive weight, gender, and insulin resistance were evaluated to explain this difference, but research suggests that underlying factors related to Latino or non-Latino background, possibly genetic and immune differences, may be affecting the response to HCV infection and treatment. However, more research is needed on the effectiveness of peginterferon and ribavirin in Latino subjects with HCV, and with combined and human immunodeficiency virus (HIV) co-infection.

Objectives:

- To evaluate the safety, effectiveness, and viral response of peginterferon alfa-2a and ribavirin therapy for chronic hepatitis C in Latino participants with and without HIV co-infection.

This is an observational study. The observed treatment is received and managed through their primary care.

DETAILED DESCRIPTION:
Hepatitis C is a major health problem affecting 100- 300 million individuals worldwide. Chronic hepatitis C virus (HCV) infection leads to cirrhosis in approximately 20% of subjects over a period of 1-20 years. Hepatitis C is now the most common indication for liver transplantation in the United States. infection occurs in one-third of all HIV-infected individuals, and the natural history among HIV-1 infected individuals demonstrates higher levels of HCV viremia, faster rates of progression and cirrhosis. There have been very few studies addressing the lower therapeutic response rates in minorities outside of African Americans. A recent study showed that Latino white subjects respond less effectively (34%) than non Latino white subjects (49%) given the same treatment even after adjusting for various important factors. As the current landscape for treatment of HCV changes, it would be important to evaluate factors responsible for therapeutic response in Latino patients.

This is a study to address the genetic, epigenetic, and proteomic expression during therapy for chronic hepatitis C in Latino participants with and without HIV co-infection. One hundred Latino participants who have evidence of chronic hepatitis C with and without HIV who are receiving treatment for HCV will be enrolled. The results of this study will enable us to explore reasons for the differential therapeutic response rates with Hepatitis C treatment in Latino participants with and without HIV coinfection.

ELIGIBILITY:
* INCLUSION CRITERIA:

A subject must satisfy all of the following criteria to be eligible to participate in this study:

1. Latino ethnicity. Latino ethnic background will be defined as a geographic, historical, and cultural heritage shared among persons from Spanish-speaking countries in South and Central America, Mexico, and the Caribbean. Both parents and all grandparents of the participant have to be Latino, with Spanish as the primary language. Participants have to be white; native aboriginal Indians, Asians, and blacks will be excluded.
2. Age greater than or equal to 18 years.
3. Documentation of hepatitis C infection by demonstration of a positive test for hepatitis C antibody and HCV RNA level of greater than or equal to 2,000 IU/mL.
4. Documentation of HIV-1 infection in the second group of co-infected participants by a licensed enzyme-linked immunosorbent assay and confirmed by a Western blot or by HIV polymerase chain reaction positive.
5. Participants with HIV: CD4+ cell counts greater than or equal to 100 cells/mm(3) or CD4+ cell percentage greater than or equal to 14%.
6. Ability to provide informed consent and willingness to comply with the study requirements, storage of blood samples and clinic policies.
7. Participants must have a primary care physician managing medical problems.
8. For HIV infected participants, care provided by a primary physician must be consistent with the current DHHS guidelines. For those on therapy, HAART will be provided by their physician.
9. Willing to undergo genetic testing
10. About to start HCV treatment (with or without direct acting agents DAAs)

EXCLUSION CRITERIA:

A subject will be ineligible to participate in this study if any of the following criteria are met:

1. Unable to comply with research study visits
2. Have any condition that the investigator considers a contraindication to study participation.
3. Pregnant or breastfeeding women.
4. Patients with poor venous access

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: latino with or without HIV infection undergoing Hepatitis C treatment
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shyamasundaran Kottilil, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Seeff LB, Hoofnagle JH. Appendix: The National Institutes of Health Consensus Development Conference Management of Hepatitis C 2002. Clin Liver Dis. 2003 Feb;7(1):261-87. doi: 10.1016/s1089-3261(02)00078-8. PMID 12691470
- [Background] Engels EA, Chatterjee N, Cerhan JR, Davis S, Cozen W, Severson RK, Whitby D, Colt JS, Hartge P. Hepatitis C virus infection and non-Hodgkin lymphoma: results of the NCI-SEER multi-center case-control study. Int J Cancer. 2004 Aug 10;111(1):76-80. doi: 10.1002/ijc.20021. PMID 15185346
- [Background] Poynard T, Bedossa P, Opolon P. Natural history of liver fibrosis progression in patients with chronic hepatitis C. The OBSVIRC, METAVIR, CLINIVIR, and DOSVIRC groups. Lancet. 1997 Mar 22;349(9055):825-32. doi: 10.1016/s0140-6736(96)07642-8. PMID 9121257

RESULTS

PARTICIPANT FLOW:
Groups:
- PegIFN and Ribavirin: Latino Patients with hepatitis C receiving weekly pegIFN and ribavirin.
  This is an observational study. The observed treatment is received and managed through their primary care.
Period: Overall Study
Arm/Group | PegIFN and Ribavirin
Started | 10
Completed | 4
Not Completed | 6
Not completed — Lack of Efficacy | 4
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: LATINO PARTICIPANTS WITH hepatitis C
Groups:
- Standard: HCV INFECTED LATINO ARTICIPANTS
Arm/Group | Standard
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 10

OUTCOME MEASURES:

1. Primary Outcome: Median Log Change in HCV RNA Levels on Day 7
Description: The primary end point of this study is the the log change in HCV RNA levels on Day 7
Time Frame: first 7 days
Measure: Median (Inter-Quartile Range); unit: log IU/mL
Arm/Group | Hepatitis C
Number analyzed (Participants) | 10
log IU/mL | NA [NA to NA] — Due to the change in the standard of care treatment of HCV, it became difficult to recruit patients to receive IFN based therapy with the prospects of IFN free treatment being available sooner. Numbers are insufficient to generate results.

ADVERSE EVENTS:
Groups:
- Standard: Patients receiving weekly peg interferon and ribavirin for hCV treatment were studied This is an observational study. The observed treatment is received and managed through their primary care.
Arm/Group | Standard
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
Early termination due to small numbers of subjects enrolled as the options for HCV treatment changed significantly since the start of the study planning.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No